CLINICAL TRIAL: NCT00416728
Title: An Open-Label, Randomized, Two-Treatment, Two Period Crossover, Single-Dose Study to Determine the Relative Bioavailability of Fixed Combination of Final Market Image (FMI) Aliskiren/Valsartan 150/80 mg Tablets and the Free Combination of Aliskiren 150 mg and Valsartan 80 mg in Healthy Subjects
Brief Title: Bioavailability of Aliskiren and Valsartan as a Single Tablet vs. the Same Doses of the Two Drugs Given Separately to Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CSPV100A2102
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: Aliskiren , Valsartan , bioavailability, hypertension; Healthy male and female subjects
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Valsartan

INTERVENTIONS:
Drug: Aliskiren
Drug: Valsartan

SUMMARY:
This study will assess the bioavailability of aliskiren and valsartan as a single tablet compared to the same doses of the two drugs given as two separate tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects 18 to 45 years (inclusive) of age in good health as determined by past medical history, physical examination, vital signs assessments, electrocardiogram, and laboratory tests at screening and baseline..
* Female subjects of child bearing potential must be using a double-barrier local contraception i.e. intra-uterine device plus condom, or spermicidal gel plus condom for at least 3 months prior to Study start or postmenopausal females must have had no regular menstrual bleeding for at least 1 year prior to inclusion (Menopause will be confirmed by a plasma FSH level of >40 IU/L) or female subjects must have been surgically sterilized at least 6 months prior to screening with supportive clinical documentation.

and all female subjects must have negative pregnancy results at screening and each baseline (regardless of reported reproductive status).

* Body mass index (BMI) must be 18 - 30 kg/m2 (inclusive) and subjects must weigh at least 50 kg.
* Vital signs should be within the following ranges: oral body temperature between 35.0-37.5 °C, systolic blood pressure, 90-140 mm Hg, diastolic blood pressure, 50-90 mm Hg, pulse rate, 40 - 90 beats per minute (bpm)

Exclusion Criteria:

* Smokers (use of tobacco products within the previous 3 months). Smokers will be defined who reports tobacco use or has a urine cotinine value of ≥ 300 ng/mL.
* Use of any prescription drugs within 4 weeks prior dosing, or over-the-counter (OTC) medication (vitamins, herbal supplements, dietary supplements) within 2 weeks prior to dosing. Acetominophen is acceptable, with supportive clinical documentation..
* Participation in any clinical investigation within a minimum of 4 weeks prior to dosing (or longer if local regulations apply).
* Significant illness within the 2 weeks prior to dosing.
* Lactating and breast feeding females.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Start 2006-11

PRIMARY OUTCOMES:
The relative bioavailability of the fixed dose combination of aliskiren/valsartan versus the free combination of aliskiren and valsartan via PK samples at pre-determined time points from pre-dose to 96 hours post-dose .

SECONDARY OUTCOMES:
To characterize the fixed dose combination of aliskiren/valsartan via PK samples at pre-determined time points.
The safety and tolerability of a single oral dose of a fixed and free combination aliskiren/valsartan.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States